CLINICAL TRIAL: NCT04479202
Title: The Effect of Berberine on Intestinal Function and Inflammatory Mediators in Severe Patients With Covid-19
Acronym: BOIFIM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Berberine treats COVID-19; XJ2020005101 (Other Grant/Funding Number: The fundamental Resrarch Funds for the Central Universities)
Record Dates: First submitted 2020-05-13; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-05

CONDITIONS: Berberine; COVID-19
Keywords: Gastrointestinal function; inflammatory biomarkers; Organ function
MeSH Terms: conditions — COVID-19 | interventions — Berberine; Bentonite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- berberine group (B group) (Experimental): Patients in the B group were given berberine hydrochloride tables 0.3g tid orally or tube feed daily, until the 14th day of the study. Other treatments include general support therapy, oxygen therapy, antiviral drugs, in combination with antibiotics and small doses of glucocorticoids if necessary, nutritional and organ function support.
  Interventions: Drug: Berberine
- control group (C group) (Sham Comparator): Patients in the C group were given montmorilonite orally if they presence of diarrhea. The other treatments were the same as in B group.
  Interventions: Drug: Montmorrillonite

INTERVENTIONS:
Drug: Berberine — Patients in the intervention group received berberine daily, regardless of gastrointestinal symptoms.If the patient has a serious drug-related adverse event, the drug will be discontinued and the patient will be excluded from the study.
  Other Names: Berberine Hydrochloride Tablets
  Arms: berberine group (B group)
Drug: Montmorrillonite — Patients in the control group were routinely not given special treatment.However, if the patient has diarrhea symptoms, montmorillonite powder should be given orally.
  Other Names: Montmorrillonite Powder
  Arms: control group (C group)

SUMMARY:
Coronavirus disease 2019 (COVID-19) rapidly spread across China and throughout the world, causing hundreds of thousands died. Studies had shown that "cytokine storms" and subsequent multiple organ dysfunction (MODS) are important causes for disease progression and death in patients with COVID-19. Similar to SARS-CoV infection, SARS-CoV-2 would infect humans via binding of S-protein to angiotensin-converting enzyme 2 (ACE2), a host cell receptor, and the S protein is activated and cleaved by cellular transmembrane serine proteases, allowing the virus to release fusion peptides for membrane fusion. In addition to the lungs, ACE2 is also highly expressed in the esophagus, small intestine and colon, suggesting that the gut might also be an important target organ for SARS-CoV-2. About 8-16% of severe pneumonia cases confirmed with SARS-CoV-2 infection developed gastrointestinal symptoms such as abdominal pain, vomiting, and diarrhea. Moreover, the stool of patient with COVID-19 also positive by real-time reverse-transcriptase-polymerase-chain-reaction (rRT-PCR) assay. Furthermore, elevated faecal calprotectin was observed in patients with COVID-19 suggested an inflammatory response in the gut, which was significantly correlated with IL-6. For severe and critical cases, control "cytokine storms" and maintain intestinal microenvironment balance have been included into the Diagnosis and Treatment Guideline of patients with COVID-19 (Edition 7). Berberine is a quaternary ammonium alkaloid isolated from rhizoma coptidis. It is often used in treatment of infectious diarrhea by bacteriostasis and inhibition of intestinal gland secretion. Berberine has also been found to have a role in intestinal immune regulation, inhibiting both AP-1 and NF- B, the key factors in cell signal transduction, and reducing the inflammatory response. Investigators conducted a prospective randomized controlled clinical trial to investigate the effects of berberine on intestinal function, serum concentrations of the inflammatory biomarkers, and organ function in severe patients with SARS-CoV-2 infection.

DETAILED DESCRIPTION:
Patients aged 18-80 years who confirmed with COVID-19 and classified as severe were enrolled in the study, and then separated randomly into two groups: a berberine group (B group) and a control group (C group). The diagnostic criteria for severe cases are in accordance with the Diagnosis and Treatment Guideline of patients with COVID-19 issued by the National Health Commission of the People's Republic of China (Edition 7). In general, patients diagnosed with COVID-19 pneumonia must also meet any of the following criteria: appears shortness of breath, respiratory rate (RR) ≥ 30 times/min; SPO2 ≤ 93% at rest; the ratio of partial oxygen pressure of arterial blood (PaO2) to oxygen absorption concentration (FiO2) ≤ 300mmHg (1mmHg=0.133KPa); pulmonary imaging showed the lesion progression >50% within 24-48 hours. All enrolled patients were given general support therapy, oxygen therapy, antiviral drugs, in combination with antibiotics and small doses of glucocorticoids if necessary, nutritional and organ function support. Patients in the berberine group (B group) were given berberine 0.3g tid orally or tube feed daily, while patients in the control group (C group) were given montmorilonite orally if they presence of diarrhea. The duration of the study intervention was 14 days and followed up to discharge. Investigators record general information about patients at admission, including age, gender, age, exposure history, time from onset of symptoms to hospital, APACHE II score, the presentation of X-ray, comorbidity, mechanical ventilation, fever or not,gastrointestinal symptoms. Investigators also evaluate the gastrointestinal function daily,including gastrointestinal symptoms (nausea, vomiting, abdominal pain, abdominal distension or diarrhoea), frequency of diarrhea, the characteristics of stool (Bristol scal). Peripheral blood are collected on day 1,3, 7 and 14 after admission to determine the level of interleukin-6 (IL-6), interleukin-1β (IL-1β), interleukin-10 (IL-10) and tumor necrosis factor (TNF-α). Laboratory tests are also performed to evaluate leucocyte, c-reactive protein (CRP), and procalcitonin (PCT) levels at the same time. Glutamate transaminase (ALT), glutamate transaminase (AST), urea nitrogen (Bun), creatinine, prothrombin time (PT), partially activated prothrombin time (APTT), and Sequential Organ Failure Assessment (SOFA) score are used to evaluate organ function on day 1,3, 7 and 14 after admission. Investigators also record the adverse events associated with the drug, length of stay and the prognosis at discharge. The patients are blinded to the group allocation. Two physicians are responsible for data processing, one is responsible for recording and collecting, and the other is responsible for checking, and they are all blind to the research.

ELIGIBILITY:
Inclusion Criteria:

* Patients confirmed with COVID-19 and classified as severe

Exclusion Criteria:

* inflammatory bowel disease;
* have other sources of infection;
* death is anticipate within 72 hours;
* participated in other clinical trials;
* pregnant or lactating women;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-02-08 (Actual); Primary Completion 2020-04-18 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Changes in diarrhea frequency and Bristol Stool Scale | daily, from date of randomization until the date of discharge or date of death from any cause, assessed up to 2 weeks.
  Including diarrhea in times/day, Bristol Stool Scale (the minimum 1 and maximum 7, a higher scores mean a worse outcome) and whether patient has any one of gastrointestinal symptoms (nausea, vomiting, abdominal pain, abdominal distension or diarrhoea).

SECONDARY OUTCOMES:
IL-6 (ng/ml) | baseline (at admission), day 3,7 and14 after admission or until the date of discharge or date of death from any cause
  evaluate inflammatory response, blood sample collected at 6:00am
IL-10（ng/ml） | baseline (at admission), day 3,7 and14 after admission or until the date of discharge or date of death from any cause
  evaluate inflammatory response, blood sample collected at 6:00am
IL-1β (ng/ml) | baseline (at admission), day 3,7 and14 after admission or until the date of discharge or date of death from any cause
  evaluate inflammatory response, blood sample collected at 6:00am
TNF-α (pg/ml) | baseline (at admission), day 3,7 and14 after admission or until the date of discharge or date of death from any cause
  evaluate inflammatory response, blood sample collected at 6:00am
leukocyte count (10^9/l) | baseline (at admission), day 3,7 and14 after admission or until the date of discharge or date of death from any cause
  evaluate inflammatory response, blood sample collected at 6:00am
c reactive protein (mg/l) | baseline (at admission), day 3,7 and14 after admission or until the date of discharge or date of death from any cause
  evaluate inflammatory response, blood sample collected at 6:00am
procalcitonin (ng/ml) | baseline (at admission), day 3,7 and14 after admission or until the date of discharge or date of death from any cause
  evaluate inflammatory response, blood sample collected at 6:00am

OTHER OUTCOMES:
Sequential Organ Failure Assessment (SOFA) score | baseline (at admission), day 3, 7 and 14 after admission or until the date of discharge or date of death from any cause
  evaluate the severity of the disease(the minimum 0 and maximum 24, a higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Wenkui Yu, M.D., Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
We have other articles about covid-19 yet to be published

REFERENCES:
- [Result] Effenberger M, Grabherr F, Mayr L, Schwaerzler J, Nairz M, Seifert M, Hilbe R, Seiwald S, Scholl-Buergi S, Fritsche G, Bellmann-Weiler R, Weiss G, Muller T, Adolph TE, Tilg H. Faecal calprotectin indicates intestinal inflammation in COVID-19. Gut. 2020 Aug;69(8):1543-1544. doi: 10.1136/gutjnl-2020-321388. Epub 2020 Apr 20. No abstract available. PMID 32312790
- [Result] Jin X, Lian JS, Hu JH, Gao J, Zheng L, Zhang YM, Hao SR, Jia HY, Cai H, Zhang XL, Yu GD, Xu KJ, Wang XY, Gu JQ, Zhang SY, Ye CY, Jin CL, Lu YF, Yu X, Yu XP, Huang JR, Xu KL, Ni Q, Yu CB, Zhu B, Li YT, Liu J, Zhao H, Zhang X, Yu L, Guo YZ, Su JW, Tao JJ, Lang GJ, Wu XX, Wu WR, Qv TT, Xiang DR, Yi P, Shi D, Chen Y, Ren Y, Qiu YQ, Li LJ, Sheng J, Yang Y. Epidemiological, clinical and virological characteristics of 74 cases of coronavirus-infected disease 2019 (COVID-19) with gastrointestinal symptoms. Gut. 2020 Jun;69(6):1002-1009. doi: 10.1136/gutjnl-2020-320926. Epub 2020 Mar 24. PMID 32213556
- [Result] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076